CLINICAL TRIAL: NCT06886945
Title: An Integrated Neurophysiological Approach Toward the Early Detection of Psychiatric Disorders
Status: Recruiting | Type: Observational
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-SCZ-EXP1
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia Disorders
Keywords: Schizophrenia; Audio-Visual Integration; Temporal Binding Windows; Signal Detection Theory; Schizotypal Personality
MeSH Terms: conditions — Schizophrenia; Schizotypal Personality Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- SCZ: Patients diagnosed with schizophrenia spectrum disorders
  Interventions: Other: Audio-Visual Perceptual Tasks
- LST: Healthy individuals displaying low schizotypal traits
  Interventions: Other: Audio-Visual Perceptual Tasks
- HST: Healthy individuals displaying high schizotypal traits
  Interventions: Other: Audio-Visual Perceptual Tasks

INTERVENTIONS:
Other: Audio-Visual Perceptual Tasks — Around 75 participants will be recruited for this study (25 per each group), and asked to perform two distinct audiovisual tasks (run via Matlab-based automated routines, and presented using a CRT monitor and a pair of loudspeakers) :
  1. TOJ task, in which a white flashing dot, and a basic auditory stimulus, will be presented in close temporal proximity at several stimulus onset asynchronies (SOAs, from 30 to 540 ms in steps of 30 ms), with participants asked to report ( after each trial), which stimulus occurred first (task duration estimate: 25 minutes, 30 trials per each SOA)
  2. A modified version of the SIFI (mSIFI), in which the presentation of paired (and temporally close) auditory stimuli will be coupled with the occurrence of either 1 or 2 flashing dots, at several different SOAs (from 30 to 250 ms in steps of 10 ms), with participants asked to report (after each trial), whether they saw 1 vs 2 flashes (task duration estimate: 25 minutes, 30 trials per each SOA)

SUMMARY:
Schizophrenia (SCZ) is a severe neuropsychiatric disorder characterized by cognitive decline, social withdrawal, and positive symptoms such as hallucinations and delusions. Research suggests that SCZ and schizotypy exist along a continuum, with shared structural and behavioral abnormalities, the latter of which encompass the sensory and perceptual domain, often in the form of altered multisensory integration, as seen in tasks like the Sound-Induced Flash Illusion (SIFI). Individuals with schizotypal traits or SCZ show enlarged temporal binding windows (TBW) of cross-modal integration, affecting perceptual accuracy and multisensory judgments. However, whether these deficits stem from overactive top-down modulation or weakened bottom-up sensory precision remains unclear.

The current study seeks to address these questions, by asking participants (healthy individuals screened as for their schizotypal traits, and patients suffering from SCZ) to complete a modified version of the SIFI, as well as an audiovisual temporal order judgment (TOJ) task. Cross-modal performance will be assessed via signal detection theory (SDT) metrics and psychometric modeling to estimate individual TBWs, thereby assaying audiovisual processing abilities along the schizotypal continuum

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is among the most debilitating syndromes within the neuropsychiatric domain, with patients suffering from this condition displaying a rich nosographic characterization. Besides, anhedonia, social withdrawal, and a progressive cognitive decline, positive manifestations such as delusions and hallucinations are perhaps the hallmark symptomatological features underlying this disorder. Notably, prodromal stages that entail subclinical cognitive and/or psychotic symptoms have often been shown to anticipate SCZ onset, corroborating a dimensional approach toward the understanding of such psychiatric disorder. Indeed, it has been proposed that schizotypal traits exist within the general population and that schizotypy and SCZ may correspond to quantitative poles within the same continuum, with the former (i.e., individuals characterized with high schizotypal traits, HST) including subjects displaying many SCZ-related subthreshold clinical signs, and thus, more likely to develop the latter. However, no reliable biomarker to early detect such psychosis-prone individuals has been so far, leaving clinicians without pre-emptive policies toward risk mitigation.

It should be nonetheless highlighted that both demeaned microstructural and white matter integrity have been reported in schizotypy and SCZ alike, the magnitude of which predicting the severity of positive symptoms at the individual level. Given the pivotal role these neuroanatomical features play in relaying electrical signals across the brain, it is not surprising that SCZ patients, as well as HST individuals, oftentimes exhibit aberrant oscillatory dynamics within the low-frequency ranges, such as in the alpha band (7-13 Hz). These brain oscillations are the dominant rhythm in both the resting and active brain. As such, they have been found to subserve many functions closely tied to sensory processing. Among multifold operational features these rhythms appear to be endowed with, their occipital cycling speed (i.e., individual alpha frequency peak, also known as IAF) has been recently associated with the efficiency by which sensory information is integrated or segregated, according to the task at hand . In agreement with the discrete sampling hypothesis of perception, the faster (or slower) these rhythms oscillate, the higher (or lower) the observers' visual sampling rate and their perceptual or cognitive accuracy.

Of note, this electrocortical index bears trait-like features that have been shown to parametrize perceptual performance, especially in multisensory contexts.

For instance, the propensity to report an illusory percept in audiovisual tasks such as the Sound-Induced Flash Illusion (SIFI) was found to negatively correlate with the IAF as recorded from occipital loci: the slower the IAF, the greater the number of illusory percepts and vice-versa. These results align with pieces of research showing a critical contribution of alpha oscillatory speed when individuals are asked to perform cross-modal simultaneity judgments and visuo-tactile tasks as well. Intriguingly, evidence for a tie between the IAF and multisensory temporal binding windows (TBW) has been further reinvigorated by data showing slower IAFs in patients suffering from schizophrenia or displaying schizotypal traits. Namely, those clinical and subclinical populations performing poorly at the SIFI, and, more broadly, multisensory paradigms, due to enlarged TBWs.

As for the neurocomputational mechanics subsiding this intricate pattern of alterations, it remains a matter of debate whether they might be driven either by an over-exploitation of auditory-relayed priors, or poor bottom-up sensory processing. Indeed, although alterations in sensory integration/segregation are a core hallmark of SCZ, it is not entirely clear whether such behavioral and cognitive impairments might be due to defective sensory processing (i.e. poor sensory input due to reduced feedforward connectivity), or aberrant perceptual bias mechanisms (i.e. disproportionately high top-down signaling), and to which extent they may be present at prodromal stages of the disease. To this aim, we will therefore investigate the performance of SCZ patients, and individuals displaying either high (HST) or low (LST) schizotypal traits, in a series of tasks relying on multisensory interaction. We will do so by implementing signal detection theory (SDT) matched with logistic fitting, to clarify at a finer-grained level whether alterations in multisensory processes can be accounted for by deficits at the level of sensory input (d'), top-down control (c), or both.

ELIGIBILITY:
Inclusion Criteria (all participants):

* Normal hearing
* Normal or corrected-to-normal vision

Inclusion Criteria (patients):

* Clinical diagnosis of schizophrenia spectrum disorder (according to DSM-5)
* IQ > 70

Exclusion Criteria (all participants):

* Anamnesis or evidence of any central nervous system alteration

Exclusion Criteria (patients)

* Current major physical illness
* Drug dependency/abuse over the last 6 months
* Unstable pharmacological therapy
* Comorbidities with other major psychiatric disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants assigned either to the low (LST) or high (HST) schizotypal group will be recruited from the general population, after being screened for their schizotypal traits via the Schizotypal Personality Questionnaire (SPQ, Raine, 1991). Individuals with SPQ scores falling within the first and last quintile of the overall SPQ scores distribution will then be recruited and assigned, respectively, to the LST and HST groups.
  SCZ patients will be recruited via the Psychiatric Unit of IRCCS Centro San Giovanni di Dio Fatebenefratelli
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Temporal Binding Window (TBW) length | Right after tasks completion
  The temporal binding window (TBW) is a psychophysical construct that reflects an observer's tolerance for temporal asynchrony-a "window" of time within which multisensory stimuli are likely to be perceptually bound or integrated. As such, it serves as a proxy for cross-modal performance.
  In both tasks, individual TBWs will be estimated for each participant by fitting gaussian and sigmoidal logistic functions to error rates (i.e., inverse accuracy) and perceptual sensitivity metrics (i.e., d', as computed combining hits and flase alarms according to signal detection theory), respectively, across the asynchrony space (e.g., at each SOA). The width (e.g., standard deviation) of the gaussian function and the inflection point (e.g., midpoint) of the sigmoidal curve will be then derived on a participant-by-participant basis, serving as behavioral indices of TBW span (in milliseconds) for further statistical analyses and comparison between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided